CLINICAL TRIAL: NCT05546177
Title: Effect Of Instrumented Assisted Soft Tissue Mobilization On Pain, Function And Proprioception In Patients With Shoulder Impingement Syndrome. A Randomised Controlled Trial
Brief Title: Effect Of Instrumented Assisted Soft Tissue Mobilization On Pain, Function And Proprioception In Patients With Shoulder Impingement Syndrome
Acronym: SIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nabil Mahmoud Ismail Abdel-Aal, Nabil mahmoud ismail, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: p.t.REC/012/002833
Record Dates: First submitted 2022-09-15; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Shoulder Impingement
Keywords: instrumented assisted soft tissue mobilization; shoulder impingement syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Intervention Model Description: instruments assisted soft tissue mobilization and traditional therapy
Who Masked: Investigator, Outcomes Assessor
Masking Description: opaque sealed envelop
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- instrumented assisted soft tissue mobilization (Experimental): the patients will receive instrumented assisted soft tissue mobilization three times a week for eight weeks
  Interventions: Other: instrumented assisted soft tissue mobilization; Other: traditional therapy
- traditional therapy (Active Comparator): the patients will receive traditional therapy three times a week for eight weeks
  Interventions: Other: traditional therapy

INTERVENTIONS:
Other: instrumented assisted soft tissue mobilization — The subject will be treated with instrumented assisted soft tissue mobilization, applied to the upper and lower fibers of Pectoral, Trapezius (upper, middle and lower), Rhomboids major , Rhomboids minor, Teres minor, Teres major, and Latissimus dorsi muscles. The IASTM technique was performed for 20 seconds parallel to the muscle fibers followed by 20 seconds perpendicular to the muscle fibers of each one of the selected muscle
  Arms: instrumented assisted soft tissue mobilization
Other: traditional therapy — the patients will receive Transcutaneous electrical nerve stimulation (TENS) to manage the pain,Ultrasound , Exercise including (Range of motion exercises, stretching exercises, and strengthening exercises (Scapular stabilization exercises and rotator cuff strengthening exercises)

SUMMARY:
this study will be conducted to investigate instrumented Assisted Soft Tissue Mobilization On Pain, Function And Proprioception In Patients With Shoulder Impingement Syndrome

DETAILED DESCRIPTION:
Shoulder impingement is a clinical syndrome in which soft tissues become painfully entrapped in the area of the shoulder joint. Patients present with pain on elevating the arm or when lying on the affected side. Shoulder pain is the third most common musculoskeletal complaint in orthopedic practice, and impingement syndrome is one of the more common underlying diagnoses. On the pathophysiological level, it can have various functional, degenerative, and mechanical causes. The impingement hypothesis assumes a pathophysiological mechanism in which different structures of the shoulder joint come into mechanical conflict. The decision to treat conservatively or surgically is generally made on the basis of the duration and severity of pain, the degree of functional disturbance, and the extent of structural damage. The goal of treatment is to restore pain-free and powerful movement of the shoulder joint.Instrument-assisted soft tissue mobilization (IASTM) is a popular treatment for myofascial restriction which is applied using specially designed instruments to provide a mobilizing effect to soft tissue (e.g., scar tissue and myofascial adhesion) to decrease pain and improve range of motion (ROM) and function. eighty patients will be allocated randomly into two equal groups; the experimental one will receive IASTM and the control will receive traditional therapy for eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with impingement syndrome from both genders.
* Age range from 25-40 years
* Body mass index 18.5-24.9 kg/m2
* Subjects are non-smokers.
* Shoulder impingement symptoms lasting at least 6 weeks

Exclusion Criteria:

1. Hand truma, present pain or other kinds of complaints in the hand area.
2. History of deformities, fractures, or surgery of the tested upper extremity joints affecting hand grip strength within the last 6 months.
3. Presence of cardiopulmonary, hormonal disorder, central or peripheral neurological deficits or any condition that can influence the results.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-09-25 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
pain intensity | up to eight weeks
  pain will be measured by visual analogue scale. It is a vertical or horizontal 100 mm line graduated by different levels of pain, starting from 0 (no pain) till 100 (worst pain)
shoulder disability | up to eight weeks
  The Arabic version of Disabilities of arm, shoulder, and hand (DASH) will be used for assessing shoulder function. DASH questionnaire includes 30 items with score from 0 to 100. A score of 0 represents no disability, while a score of 100 represents the most sever.

SECONDARY OUTCOMES:
shoulder range of motion | up to eight weeks
  inclinometer will be used to assess shoulder range of motion.
shoulder proprioception | up to eight weeks
  inclinometer will be used to assess shoulder proprioception
rounded shoulder | up to eight weeks
  tape measure will be used to assess the rounded shoulder